CLINICAL TRIAL: NCT00395343
Title: A Phase III, Multicenter, Randomized, Double-Blind Clinical Trial to Study the Safety and Efficacy of the Addition of Sitagliptin (MK0431) to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Insulin Therapy (Alone or In Combination With Metformin)
Brief Title: Sitagliptin Added-on to Insulin Study (0431-051)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-051; MK0431-051; 2006_532
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2009-10-23 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): sitagliptin
  Interventions: Drug: sitagliptin phosphate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator : placebo (unspecified)

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin 100 mg tablet qd for a 24-wk treatment period.
  Other Names: MK0431; Januvia™
  Arms: 1
Drug: Comparator : placebo (unspecified) — sitagliptin 100 mg Pbo tablet qd for a 24-wk treatment period.
  Arms: 2

SUMMARY:
A clinical study to determine the safety and efficacy of sitagliptin in patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on insulin or insulin/metformin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Patient is poorly controlled while on insulin or insulin and metformin

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient is taking oral antidiabetic agents other than metformin during the past 3 months
* Patient is currently on treatment with daily use of pre-prandial short-acting or rapid-acting insulin

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2006-12-11 (Actual); Primary Completion 2008-10-13 (Actual); Study Completion 2008-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Vilsboll T, Rosenstock J, Yki-Jarvinen H, Cefalu WT, Chen Y, Luo E, Musser B, Andryuk PJ, Ling Y, Kaufman KD, Amatruda JM, Engel SS, Katz L. Efficacy and safety of sitagliptin when added to insulin therapy in patients with type 2 diabetes. Diabetes Obes Metab. 2010 Feb;12(2):167-77. doi: 10.1111/j.1463-1326.2009.01173.x. PMID 20092585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 29-Jan-2007 Last Patient Last Visit: 13-Oct-2008; 100 study centers worldwide
Pre-assignment Details: Patients at least 21 years of age with type 2 diabetes mellitus with inadequate glycemic control (A1C ≥7.5 and ≤11.0%) on stable-dose insulin (alone or in combination with stable-dose metformin) were eligible to enter the 24 week study. 1-week screening, followed by a 2-week single-blind placebo run-in.
Groups:
- Sitagliptin 100 mg q.d.: The Sitagliptin 100 mg q.d. (q.d. = once daily) group includes data from patients randomized to receive treatment with 100 mg oral tablets of sitagliptin once daily (blinded) in addition to ongoing treatment with insulin (pre-mixed, intermediate-acting, or long-acting) alone or in combination with open-label metformin 500 mg oral tablets (≥1500 mg/day).
- Placebo: The Placebo group includes data from patients randomized to receive treatment with a placebo of the sitagliptin 100 mg oral tablet once daily (blinded) in addition to ongoing treatment with insulin (pre-mixed, intermediate-acting, or long-acting) alone or in combination with open-label metformin 500 mg oral tablets (≥1500 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Started | 322 | 319
Completed | 281 | 283
Not Completed | 41 | 36
Not completed — Adverse Event | 13 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Physician Decision | 2 | 4
Not completed — Protocol Violation | 6 | 8
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg q.d. | Placebo | Total
Number analyzed (Participants) | 322 | 319 | 641
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.1) | 57.2 (9.3) | 57.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 150 | 315
  Male | 157 | 169 | 326
Race/Ethnicity, Customized [Number; unit: participants]
  White | 228 | 219 | 447
  Black | 21 | 23 | 44
  Asian | 55 | 61 | 116
  Other | 18 | 16 | 34
A1C (Hemoglobin A1c) [Mean (Standard Deviation); unit: Percent] | 8.7 (0.9) | 8.6 (0.9) | 8.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: A1C is measured as a percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last non-baseline observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 305 | 312
Percent | -0.59 [-0.70 to -0.48] | -0.03 [-0.14 to 0.08]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; metformin stratum (on vs. not on metformin); insulin stratum (pre-mixed vs. intermediate or long-acting); Mean Difference (Net) = -0.56, 95% CI [-0.70 to -0.42]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 310 | 313
mg/dL | -18.5 [-25.1 to -11.9] | -3.5 [-10.2 to 3.1]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; metformin stratum; insulin stratum; Mean Difference (Net) = -15.0, 95% CI [-23.4 to -6.5]

3. Secondary Outcome: Change From Baseline in 2-hour Post-meal Glucose (PMG) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 240 | 257
mg/dL | -30.9 [-40.0 to -21.8] | 5.2 [-3.6 to 13.9]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; metformin stratum; insulin stratum; Mean Difference (Net) = -36.1, 95% CI [-47.1 to -25.1]

4. Secondary Outcome: Percent Change From Baseline in Index of Static Beta-Cell Sensitivity to Glucose at Week 24
Description: Static sensitivity is a measure of the effect of glucose on beta-cell secretion and is the ratio between the insulin secretion rate and glucose concentration above the threshold level at steady state. (See Breda and Cobelli, Annals of Biomedical Engineering 29, 692-700 (2001) for more details.)
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included all patients who participated in the 10-point meal tolerance test and had a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last non-baseline observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 35 | 45
Percent | 28.4 [5.4 to 56.6] | -8.1 [-22.6 to 9.2]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.01, ANCOVA; Model terms: treatment; log-scaled baseline value; metformin stratum; insulin stratum; Geometric Mean Difference = 36.5, 95% CI [8.9 to 64.7]

5. Secondary Outcome: Percent of Patients With A1C < 7.0% at Week 24
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 305 | 312
Percent | 12.8 | 5.1
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, Logistic Regression — Based on a test of the odds ratio = 1, comparing the odds of having A1C <7.0% at Week 24 in the Sitagliptin 100 mg q.d. group vs. the Placebo group; Model terms: treatment; baseline; Metformin stratum; and insulin stratum; Odds Ratio (OR) = 3.60, 95% CI [1.89 to 6.85]

6. Secondary Outcome: Percent of Patients With A1C < 6.5% at Week 24
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 305 | 312
Percent | 2.3 | 1.9
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.584, Logistic Regression — [p-value comment as in outcome 5, analysis 1]; Model terms: treatment; baseline; Metformin stratum; and insulin stratum; Odds Ratio (OR) = 1.37, 95% CI [0.45 to 4.18] — This parameter estimate and 95% confidence interval correspond to the odds of having A1C <6.5% at Week 24 in the Sitagliptin 100 mg q.d. group vs. the Placebo group

7. Other Pre Specified Outcome: Change From Baseline in A1C at Week 24
Description: A1C in subset of patients on long-acting or intermediate-acting insulin.
  A1C is measured as a percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) included the subset of patients on long-acting or intermediate-acting insulin with a baseline value and ≥1 post-baseline value for this outcome. Data following glycemic rescue were treated as missing. For FAS patients with no data at Week 24, the last non-baseline observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Number analyzed (Participants) | 225 | 232
Percent | -0.61 [-0.73 to -0.48] | -0.04 [-0.16 to 0.08]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment; baseline; metformin stratum; insulin stratum, treatment by insulin stratum interaction; Mean Difference (Net) = -0.56, 95% CI [-0.72 to -0.40]

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg q.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 20/322 | 11/319
Other Adverse Events (participants affected / at risk) | 49/322 | 25/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg q.d. (N=322) | Placebo (N=319)
Any Cardiac disorders (Cardiac disorders) | 4 | 5
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Any Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Any Infections and Infestations (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0
Genital abscess (Infections and infestations) | 1 | 0
Perianal abscess (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Any Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Any Investigations (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Any Neoplasms Benign, Malignant and Unspecified (Incl Cysts and Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Any Nervous System Disorders (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Any Psychiatric Disorders (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Any Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Any Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Any Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 2 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Any Vascular Disorders (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg q.d. (N=322) | Placebo (N=319)
Any Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 49 | 25
Hypoglycaemia (Metabolism and nutrition disorders) | 49 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.